CLINICAL TRIAL: NCT00361049
Title: Donor Mesenchymal Stem Cell Infusion for Treatment of Graft Versus Host Disease: A Phase I Trial
Brief Title: Donor Mesenchymal Stem Cell Infusion in Treating Patients With Acute or Chronic Graft-Versus-Host Disease After Undergoing a Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Hillard M. Lazarus, M.D., Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU3Y03; P30CA043703 (NIH); CASE-CWRU-3Y03 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Cancer
Keywords: graft versus host disease; unspecified adult solid tumor, protocol specific; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage II ovarian epithelial cancer; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III ovarian epithelial cancer; stage III small lymphocytic lymphoma; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV ovarian epithelial cancer; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Neoplasms; Graft vs Host Disease; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Multiple Myeloma; Carcinoma, Ovarian Epithelial; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Testicular Neoplasms; Breast Neoplasms | interventions — Therapeutics; In Situ Hybridization, Fluorescence; Immunoenzyme Techniques; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: graft versus host disease prophylaxis/therapy — Within 72 hours after the initiation of medical therapy (e.g., corticosteroids, cyclosporine) for graft-vs-host disease, patients undergo donor MSC infusion over 10-15 minutes.
Genetic: fluorescence in situ hybridization — Tissue specimens are examined by CD45 immunohistochemistry and fluorescent in situ hybridization to detect hematopoietic and nonhematopoietic cells.
Other: immunoenzyme technique — Tissue specimens are examined by CD45 immunohistochemistry and fluorescent in situ hybridization to detect hematopoietic and nonhematopoietic cells.
Other: immunohistochemistry staining method — Tissue specimens are examined by CD45 immunohistochemistry and fluorescent in situ hybridization to detect hematopoietic and nonhematopoietic cells.
Other: laboratory biomarker analysis — Tissue specimens are examined by CD45 immunohistochemistry and fluorescent in situ hybridization to detect hematopoietic and nonhematopoietic cells.
Procedure: in vitro-treated bone marrow transplantation — Within 72 hours after the initiation of medical therapy (e.g., corticosteroids, cyclosporine) for graft-vs-host disease, patients undergo donor MSC infusion over 10-15 minutes.
Procedure: management of therapy complications — Patients will be evaluated for clinical signs and symptoms of GVHD weekly for up to 28 days.

SUMMARY:
RATIONALE: Donor mesenchymal stem cell infusion may be an effective treatment for acute or chronic graft-versus-host disease caused by a donor stem cell transplant.

PURPOSE: This phase I trial is studying the side effects and best dose of donor mesenchymal stem cells in treating patients with acute or chronic graft-versus-host disease after undergoing a donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of donor mesenchymal stem cell (MSC) infusion in patients with acute or extensive chronic graft-vs-host disease (GVHD) after undergoing HLA-identical sibling donor stem cell transplant.

Secondary

* Describe the rates of complete and partial resolution of GVHD when MSCs are used in addition to the standard GVHD therapy.
* Determine inflammatory cytokine levels, lymphocyte subsets, and donor-reactive lymphocyte numbers in blood of patients with acute GVHD prior to therapy and at 7 and 14 days post-MSC therapy.
* Determine if donor MSCs engraft in tissues inflamed by GVHD in patients who have undergone gender-mismatched transplantation.

OUTLINE: This is a multicenter, dose-escalation study of donor mesenchymal stem cells (MSC).

Within 72 hours after the initiation of medical therapy (e.g., corticosteroids, cyclosporine) for graft-vs-host disease, patients undergo donor MSC infusion over 10-15 minutes.

Cohorts of 3-6 patients receive escalating doses of donor MSCs until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Blood samples are obtained periodically and examined by immunoenzyme techniques for mixed lymphocyte reaction (as a surrogate marker for alloreactivity) and cytokine levels (TH1 [i.e., interleukin (IL)-2 and interferon-gamma], TH2 [i.e., IL-10 and IL-4], and inflammatory cytokines [i.e., tumor necrosis factor-alpha and IL-1]). Tissue specimens are examined by CD45 immunohistochemistry and fluorescent in situ hybridization to detect hematopoietic and nonhematopoietic cells.

After completion of study treatment, patients are followed periodically for 1 year.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Developed acute graft-vs-host disease (GVHD) of clinical grade II-IV or extensive chronic GVHD after undergoing HLA-identical sibling donor hematopoietic stem cell transplant for any indication, malignant or nonmalignant

  * Requires systemic immunosuppressive therapy with systemic corticosteroids (methylprednisone dose 2 mg/kg/day or equivalent) and concurrent cyclosporine or tacrolimus
* May have been enrolled on an institutional allogeneic stem cell transplant protocol using either ablative or nonmyeloablative preparative regimens
* No evidence of relapsed or progressive malignant disease at the time of GVHD

PATIENT CHARACTERISTICS:

* Not pregnant
* Negative pregnancy test
* Creatinine clearance ≥ 20 mL/min
* Oxygen saturation ≥ 90% on room air
* No severe or symptomatic restrictive or obstructive lung disease or respiratory failure requiring ventilator support
* No uncontrolled hypertension or congestive heart failure, active angina pectoris requiring the use of nitrates, myocardial infarction within the past 6 months, or major ventricular arrhythmia or cardiac failure requiring active treatment
* No significant organ dysfunction
* No active severe infections, including sepsis, pneumonia with hypoxemia, persistent bacteremia, or meningitis

  * Fever without a source is allowed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-09; Primary Completion 2009-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety | Monitored for 6 hours for infusion related toxicity. Temperature, blood pressure, pulse and O2 saturation will be measured at baseline and every 10 minutes x 2, every 30 minutes x 2, and every hour x 3.

SECONDARY OUTCOMES:
Complete and partial resolution of graft-vs-host disease (GVHD) | Patients will be evaluated for clinical signs and symptoms of GVHD weekly for up to 28 days.
Cytokine levels, lymphocyte subsets, and donor-reactive lymphocyte numbers in patients with acute GVHD | Pre-transplant, at diagnosis, 7 and 14 days after MSC infusion

CONTACTS AND LOCATIONS:
Overall Officials: Hillard M. Lazarus, MD, Principal Investigator — Ireland Cancer Center at University Hosptials Case Medical Center, Case Comprehensive Cancer Center
Locations (8):
- United States (8):
  - Geauga Regional Hospital, Cleveland, Ohio
  - Lake/University Ireland Cancer Center, Cleveland, Ohio
  - Ireland Cancer Center at University Hosptials Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University Suburban Health Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - Southwest General Health Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Cleveland, Ohio